Official Title: A Randomized Clinical Trial of 100 Units of Intradetrusor Onabotulinum Toxin A for Refractory Overactive Bladder - Is 10 Injections Less Painful Than 20 Injections?

NCT04124939 Date: 7/31/23

## Statistical Analysis - 10 vs 20 Botox Injections

Standard descriptive statistics were used to compare demographic and clinical characteristics. Frequency and percentages were reported for categorical data. Chi-square and fisher exact test for categorical variables and student t-test or Mann-Whitney U test for continuous variables were used to assess significant differences between the groups. Statistical analysis was performed on R Software.